CLINICAL TRIAL: NCT04862884
Title: A Phase 1, Single Center, Randomized, Double-blind, Placebo-controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, on the Pharmacokinetics of HRS4800 in Healthy Male Subjects
Brief Title: A Trial to Evaluate the Safety and PK Profile of HRS4800 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS4800-101
Record Dates: First submitted 2021-04-19; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: HRS4800 tablets single administration in healthy male
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS4800 tablets (Experimental)
  Interventions: Drug: HRS4800 tablets
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HRS4800 tablets — 1. Drug: HRS4800 tablets Low-dose group, single oral administration
  2. Drug: HRS4800 tablets Low-medium dose group, single oral administration
  3. Drug: HRS4800 tablets medium -dose group, single oral administration
  4. Drug: HRS4800 tablets Medium and high dose group, single oral administration
  5. Drug: HRS4800 tablets High-dose group, single oral administration
  Arms: HRS4800 tablets
Drug: placebo — 1. Drug: placebo Low-dose group, single oral administration
  2. Drug: placebo Low-medium dose group, single oral administration
  3. Drug: placebo medium -dose group, single oral administration
  4. Drug: placebo Medium and high dose group, single oral administration
  5. Drug: placebo High-dose group, single oral administration
  Arms: placebo

SUMMARY:
The study will be conducted to evaluate the safety and PK profile of HRS4800 tablets after single oral administration in different dose levels compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purposes and risks of the trial and comply with all study procedures before entering the trial, and provide signed informed consent.
2. Male aged between 18 years and 55 years at screening, inclusive.
3. Total body weight ≥50 kg at screening, and body mass index (BMI) between 19.0 and 26.0 kg/m2, inclusive.
4. Agree to take contraceptive measures and promise not to donate sperm since signing the informed consent form, to 3 months after the administration.
5. No clinically significant abnormalities in medical history, general physical examination, vital signs, laboratory tests (hematology, urinalysis, blood chemistry, coagulation function), and ECG, as determined by the investigator.

Exclusion Criteria:

1. History of severe digestive system disease or having a digestive disease currently within 3 months of screening or before first dosing, and may affect drug absorption or have safety risks.
2. Severe infections, injuries or surgeries within 3 months of screening or before first dosing, or plan to undergo any surgeries during the trial.
3. ALT, AST, ALP or total bilirubin level exceeds the upper limit of normal (ULN) during screening/baseline visits.
4. Subject's supine systolic BP is ≥140 mmHg or <90 mmHg; diastolic BP ≥90 mmHg or <60 mmHg at screening or before first dosing.
5. Positive breath alcohol test after confirmation in a repeat test during screening/baseline visits.
6. Positive drug screening tests,.
7. Whole blood donation or loss of more than 200 mL of blood within 1 month prior to dosing; or blood donation or loss of more than 400 mL of blood within 3 months prior to dosing; or received blood within 2 months prior to dosing.
8. History of allergy to the study drug or any component of it.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-03 (Estimated); Primary Completion 2021-09-03 (Estimated); Study Completion 2021-09-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Adverse Events (AEs) | 1-21 days
Proportion of Participants with Hematology, Clinical Chemistry, Urinalysis Laboratory Abnormalities | 1-21 days
Proportion of Participants with 12-lead electrocardiograms (ECG) Abnormalities | 1-21 days
Proportion of Participants with Vital Sign and Physical Examinations Abnormalities | 1-21 days

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of HRS4800, | 1-6 days
Time to Attain Maximum Observed Plasma Concentration (Tmax) of HRS4800, | 1-6 days
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC[last]) of HRS4800, | 1-6 days
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) of HRS4800 | 1-6 days
Apparent Terminal Elimination Half-Life (t1/2) of HRS4800, | 1-6 days
Elimination Rate Constant (λz, or kel) of HRS4800, | 1-6 days
Apparent Volume of Distribution (VZ/F) During Terminal Phase of HRS4800 | 1-6 days
Total HRS4800 of Cumulative Amount Excreted in Urine (Aeu) | 1-6 days
Total HRS4800 of Fraction of Dose Excreted in Urine (feu) | 1-6 days